CLINICAL TRIAL: NCT01057316
Title: Evaluation of Safety and Effectiveness of the Formula PTX Balloon-Expandable Stent for Renal Artery Stenosis
Brief Title: Formula PTX Renal Stent Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-008
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Renal Artery Stenosis
MeSH Terms: conditions — Renal Artery Obstruction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Study Group A (Experimental)
  Interventions: Device: Formula PTX Stent - Dose 1
- Study Group B (Experimental)
  Interventions: Device: Formula PTX Stent - Dose 2
- Study Group C (Experimental)
  Interventions: Device: Formula PTX Stent - Dose 3

INTERVENTIONS:
Device: Formula PTX Stent - Dose 1 — Stenting of the renal artery with a PTX-coated stent (experimental) or uncoated stent (active comparator). Groups are blinded.
  Arms: Study Group A
Device: Formula PTX Stent - Dose 2 — Stenting of the renal artery with a PTX-coated stent (experimental) or uncoated stent (active comparator). Groups are blinded.
  Arms: Study Group B
Device: Formula PTX Stent - Dose 3 — Stenting of the renal artery with a PTX-coated stent (experimental) or uncoated stent (active comparator). Groups are blinded.
  Arms: Study Group C

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the PTX-coating on the Formula PTX Balloon-Expandable Stent in treatment of renal artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* renal artery stenosis
* appropriate size and location of the lesion

Exclusion Criteria:

* pregnant or breast feeding
* failure or inability to give informed consent
* simultaneously participating in another drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2014-01 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Percent Diameter Stenosis of the Treated Renal Artery | 9 months

CONTACTS AND LOCATIONS:
Locations (12):
- Czechia (2):
  - University Hospital Ostrava, Ostrava-Poruba
  - Institute for Clinical and Experimental Medicine, Prague
- Hopital Europeen Georges Pomidou, Paris, France
- Germany (6):
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Krankenhaus Neu-Bethlehem, Göttingen
  - Uniklinik Heidelberg, Heidelberg
  - Universitatsklinikum Leipzig AoR, Leipzig
  - St. Bonifatius Hospital, Lingen
  - Klinik Dr. Hancken im Elbe Klinikum Stade, Stade
- United Kingdom (3):
  - Royal Sussex County Hospital, Brighton
  - Kent & Canterbury Hospital, Canterbury
  - St. Mary's Hospital, London